CLINICAL TRIAL: NCT06814652
Title: The Outcome of CYP2D6 Polymorphism on Tramadol Analgesia in Postpartum Patients in Erbil
Brief Title: The Impact of CYP2D6 Polymorphism on Tramadol Pharmacodynamics
Status: Active, not recruiting | Type: Observational
Sponsor: Elweyia Maternity Teaching Hospital (Other)
Responsible Party: Principal Investigator, Shaymaa Faruq Hamadameen, Research Investigator, Elweyia Maternity Teaching Hospital
Other Study IDs: ElweyiaMTH
Record Dates: First submitted 2025-01-28; First posted 2025-02-07 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Post-cesarean Pain; CYP2D6 Polymorphism; Tramadol Resistance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples With DNA — 2 ml of whole blood was collected in EDTA tube
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- post-cesarean patients: All of these patients were planned to undergo elective cesarean surgery and receive postpartum management for twenty-four hours at the Erbil Maternity and Childbirth Hospital. Consent was taken from each patient prior to the enrollment into the study. Their age ranged between 21-42 years. Patients received one dose of tramadol drug (100mg/2ml of Trodon® Hemofarm) intravenously for management of postpartum pain after gaining back their pain sensation.
  Interventions: Drug: Trodon® Hemofarm

INTERVENTIONS:
Drug: Trodon® Hemofarm — Consent was taken from each patient prior to the enrollment into the study during the first interview and 2 ml of blood was withdrawal for the CYP2D6 genotyping. After the cesarean section surgery, each patient received one dose of 100mg/2ml Trodon® Hemofarm for treating the postpartum pain and the patients were monitored for 24 hours. Follow-up was performed for each enrolled patient in which the VAS score, blood pressure, heart rate, oxygen saturation and any new effects after 1 hour, 6 hours of tramadol administration were recorded. In addition, after 24 hours evaluations for nocturnal pain, dietary state and bowel movement were performed.

SUMMARY:
CYP2D6 is an enzyme involved in the hepatic metabolism of many clinically important drugs: antiarrhythmics, antidepressants, antipsychotics, β-blockers, and analgesics such as tramadol and codeine. CYP2D6 is highly polymorphic and significant interindividual variability has been observed worldwide. This study aims to investigate the distribution of CYP2D6 polymorphisms among post-cesarean female patients in Erbil city, Iraq. The findings of this study may indicate the presence of CYP2D6 gene variants among the Kurdish female population in Erbil, which could contribute to tramadol analgesic failure or exaggerated adverse effects. This study could also serve as a foundation for further pharmacogenetic research, individualizing treatments and targeting a larger sample size in the future.

ELIGIBILITY:
Inclusion Criteria:

* Female patients aged between 18-56 years old
* Patients who undergo cesarean section surgery
* Patients receive tramadol drug for postpartum pain management

Exclusion Criteria:

* Patients with any history of severe renal, liver, respiratory diseases and/or seizures
* Patients with history of psychiatric disorders or unable to provide consent
* Patients with complicated surgeries or neonatal distress or unable to perform the clinical assessment of pain
* Patients with history of consumption of chronic alcohol or opioid or drug abuse
* Patients with history of known allergy to tramadol

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — female patients who were pregnant and indicated for elective cesarean section surgery for the delivery of singleton baby.
Study Population: Pregnant patients who were indicated for elective cesarean section surgery at public hospital (Maternity Teaching hospital) located in Erbil city, Iraq were enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2024-09-22 (Actual); Primary Completion 2024-12-20 (Actual); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Visual analog scale (10 cm) | after 1 hour and 6 hours of receiving single dose of tramadol
  Visual analog scale is used for measuring pain intensity on a scale of 0 to 10, in which a score on the line is marked by each patient ranging from "no pain" to "worst pain". The pain intensity increases as the score on the scale goes up.

SECONDARY OUTCOMES:
Blood pressure (mm of Hg) | after 1 hour and 6 hours of receiving single dose of tramadol
  Blood pressure was measured by automatic blood pressure monitor (mm of Hg) after 1 hour and 6 hours of IV tramadol administration to detect any change in the blood pressure of each patient.
Heart rate (beats per minute) | after 1 hour and 6 hours of receiving single dose of tramadol
  Pulse was recorded by pulse oximetry (beats per minute) after 1 hour and 6 hours of IV tramadol administration to detect any change in the heart rate of each patient.
Oxygen saturation (SPO2%) | after 1 hour and 6 hours of receiving single dose of tramadol
  Oximetry was used (SPO2 %) for evaluating the oxygen saturation of each patient.
Nocturnal pain | after 24 hours of receiving single dose of tramadol
  Evaluation of nocturnal pain was performed for each patient by a questionnaire after 24 hours to determine pain at night and whether it has impacted on the sleeping quality of the patient.
Dietary state | after 24 hours of receiving single dose of tramadol
  Evaluation of dietary state was performed for each patient, in which the patient was asked after 24 hours to determine whether they have taken anything within the last 24 hours and if yes did they take liquid and/or solid food.
Adverse effects | after 1 hour and 6 hours of receiving single dose of tramadol for recording any adverse effects, and after 24 hours of receiving single dose of tramadol for evaluation of the bowel movement (whether the patient was constipated).
  A questionnaire was presented to each patient for recording any newly appearing effects that are noticed by the patient after 1 hour and 6 hours of receiving single dose of tramadol drug intravenously. In addition, the patient was asked after 24 hours whether they had had bowel movement within the last 24 hours (whether the patient was constipated).

CONTACTS AND LOCATIONS:
Locations (1):
- Hawler Medical University/ College of Medicine, Erbil, Iraq